CLINICAL TRIAL: NCT04742036
Title: A Phase I Open-label Study to Assess the Pharmacokinetics, Safety, and Tolerability of Capivasertib Monotherapy and in Combination With Paclitaxel in Chinese Patients With Advanced Solid Tumours.
Brief Title: Capivasertib China PK Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3614C00002
Record Dates: First submitted 2021-01-15; First posted 2021-02-05 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Advanced Solid Tumours
Keywords: Pharmacokinetics; Safety; Tolerability; Capivasertib; Chinese
MeSH Terms: interventions — capivasertib; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- capivasertib (Experimental): single-dose and multiple-dose capivasertib as monotherapy (Part A) and then in combination with paclitaxel (Part B)
  Interventions: Drug: Capivasertib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Capivasertib — Part A Cycle 0: Single dose 480 mg(3 x 160 mg tablets) on Day 1 of Cycle 0 Cycle 1 (monotherapy): 480 mg(3 x 160 mg tablets) twice daily given on an intermittent weekly dosing schedule (4 days on, 3 days off for 7 days) Part B Cycle 2 (in combination therapy with paclitaxel): 400 mg (2 x 200 mg tablets) twice daily given on an intermittent weekly dosing schedule. Patients will be dosed on Days 2 to 5 of Weeks 1, 2, and 3 followed by 1 week off-treatment within each 28-day treatment cycle. Capivasertib treatment will continue until disease progression, unacceptable toxicity or the participant requests to stop treatment.
  Other Names: AZD5363
Drug: Paclitaxel — Part B Cycle 2: Patients will receive 3 consecutive weekly infusions of 80 mg/m2 (given on Day 1 of Weeks 1, 2, and 3), followed by 1 week off-treatment within each 28-day treatment cycle.
  Paclitaxel treatment will continue for at least 6 cycles, unless the participant experiences unacceptable toxicity that is attributed directly to treatment with paclitaxel, or disease progression.

SUMMARY:
This is an open-label, 2-part Phase I study to assess the PK, safety and tolerability of capivasertib as monotherapy and in combination with paclitaxel in Chinese participants with advanced solid tumours

DETAILED DESCRIPTION:
A Phase I study is designed to assess the PK, safety and tolerability of single-dose and multiple-dose capivasertib as monotherapy (Part A) and in combination with paclitaxel (Part B) in approximately 16 Chinese participants with advanced solid tumours and to detect any differences in the PK profile between Chinese and Caucasian participants due to ethnicity. Descriptive summary will be conducted on the PK analysis set and safety analysis set.The evaluation of capivasertib PK data will be based on the PK analysis set.The assessment on safety and tolerability will be based on the safety analysis set.

ELIGIBILITY:
Key inclusion criteria

* Participants must have at least 1 lesion, not previously irradiated, that can be measured accurately at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) with computer tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements, or Lytic or mixed (lytic + sclerotic) bone lesions that can be assessed by CT or MRI in the absence of measurable disease as defined above; patients with sclerotic/osteoblastic bone lesions only in the absence of measurable disease are not eligible.
* Histologically or, where appropriate, cytologically-confirmed malignant solid tumour refractory or resistant to standard therapy and for which no suitable effective standard therapy exists
* Participants must have a life expectancy of ≥12 weeks
* Participants must be eligible for paclitaxel treatment as per local investigator assessment
* ECOG performance status 0-1
* Participants must be on a stable concomitant medication regimen, defined as no changes in medication or in dose within 2 weeks prior to start of capivasertib dosing, except for bisphosphonates, denosumab and corticosteroids, which should be stable for at least 4 weeks prior to start of capivasertib dosing

Key Exclusion criteria

* Radiotherapy with a wide field of radiation within 4 weeks before the first dose of study treatment
* Other malignancies within 5 years prior to treatment initiation (except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer)
* Participants with any ongoing toxicities (>CTCAE grade 2), with the exception of alopecia, caused by previous cancer therapy
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
* Any of the following cardiac criteria at screening:

  * Mean resting corrected QT interval (QTc) >470 msec obtained from 3 consecutive ECGs
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (eg, complete left bundle branch block, third-degree heart block)
* Clinically significant abnormalities of glucose metabolism as defined by any of the following at screening:

  * Participants with diabetes mellitus type I or diabetes mellitus type II requiring insulin treatment
  * glycosylated haemoglobin (HbA1c) ≥8.0% (63.9 mmol/mol)
* Inadequate bone marrow reserve or organ function
* Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids for at least 4 weeks prior to start of study treatment
* Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment
* Refractory nausea and vomiting, malabsorption syndrome, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection, or other condition that would preclude adequate absorption of capivasertib
* Previous allogeneic bone marrow transplant or solid organ transplant
* Evidence of dementia-altered mental status or any psychiatric condition that would prohibit understanding or rendering of informed consent
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent
* Any previous treatment with AKT, PI3K, and/or mTOR inhibitors
* Participation in another clinical study with an IP administered in the last 30 days or 5 half-lives, whichever is longer.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to 12 hours post-dose (AUC 0-12) of Capivasertib | first dose up to approximately 6 months
  AUC0-12 is defined as area under the curve from 0 to 12 hours.
Maximum plasma concentration (Cmax) of Capivasertib | first dose up to approximately 6 months
  Cmax is defined as maximum plasma concentration
terminal half-life (t1/2) of Capivasertib | first dose up to approximately 6 months
  t1/2 is defined as terminal half-life
Accumulation ratio (Rac) of Capivasertib | first dose up to approximately 6 months
  Rac is defined as accumulation ratio

SECONDARY OUTCOMES:
Safety and tolerability of drugs by assessment of AEs/SAEs | From time of signature of the ICF, through study completion, up to 17 months, and including the 30-day follow-up period after discontinuation of study drug
  Graded according to the National Cancer Institute (NCI CTCAE V5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Principal Investigator — Department of Medical Oncology, Fudan University Shanghai Cancer Center; Jian Zhang, Principal Investigator — Department of Medical Oncology, Fudan University Shanghai Cancer Center
Locations (1):
- Research Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Zhang J, Liu X, Du Y, Mu Y, Meng Y, Sun Y, Zhang L, Chen C, Cullberg M, Fan E, Hu X. A Phase I open-label study to assess the pharmacokinetics, safety, and tolerability of capivasertib alone or in combination with paclitaxel in Chinese patients with advanced solid tumors. BMC Cancer. 2025 Oct 14;25(1):1562. doi: 10.1186/s12885-025-14982-4. PMID 41088025